CLINICAL TRIAL: NCT04815395
Title: The Differential Effects of Oral and Intranasal Oxytocin on Attention Control
Brief Title: Differential Effects of Oral and Intranasal Oxytocin on Attention Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-80
Record Dates: First submitted 2021-03-22; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Healthy
Keywords: Antisaccade task; Attention control; Oxytocin; Eye-tracking
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Between-subject randomized placebo-controlled double-blind pharmacological eye-tracking design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral Oxytocin (Experimental): Oxytocin (24IU) orally
  Interventions: Drug: Oxytocin
- Intranasal Oxytocin (Experimental): Oxytocin (24IU) intranasally
  Interventions: Drug: Oxytocin
- Oral Placebo (Placebo Comparator): Placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Administration of oxytocin (24IU) orally
  Arms: Oral Oxytocin
Drug: Oxytocin — Administration of oxytocin (24IU) intranasally
  Arms: Intranasal Oxytocin
Drug: Placebo — Administration of placebo orally
  Arms: Oral Placebo

SUMMARY:
The main aim of the present study is to investigate whether oxytocin (24IU) via different routes have divergent effects on attention control in a social-emotional saccade/antisaccade eye-tracking paradigm.

DETAILED DESCRIPTION:
Previous studies have demonstrated oral and intranasal oxytocin's divergent effects on arousal rating and neural responses to emotional faces, however, it remains unclear whether different routes of oxytocin treatment would have differential effects on attention processing to social stimuli. Based on the previous registered studies (ClinicalTrials.gov ID: NCT04493515 and NCT03486925) from our group using a validated emotional anti-saccade task with social stimuli (emotional faces) and non-social stimuli (oval shape) have separately explored oral and intranasal oxytocin's modulatory effects on attention processing, the present study aims to conduct a secondary analysis of the previously acquired data to directly compare oxytocin's effects on attention control to social emotional stimuli via different routes. To this end data from subjects who underwent intranasal oxytocin administration (n = 33, NCT03486925) will be compared with data from subjects who underwent oral oxytocin or placebo administration (n = 36, or 37 respectively; NCT04493515). To further control for non-treatment related factors the intranasal placebo and oral placebo groups from the previous studies (ClinicalTrials.gov ID: NCT03486925 and NCT04493515) will be compared with respect to primary and secondary outcome measures of the trial, in particular general and emotion-specific effects on attentional control.

ELIGIBILITY:
Inclusion Criteria:

* Male, healthy participants
* Non smokers

Exclusion Criteria:

* Previous or current medical, psychiatric, neurological disorder
* Regular medication
* Use of any psychoactive substances in the 24 hours before experiment
* Contra-indications for eye-tracking data acquisition

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Differential effects of intranasal and oral oxytocin administration on saccade/antisaccade latencies towards social (facial) versus non-social (shape) stimuli | 45 minutes - 100 minutes after treatment
  Comparison between social-specific saccade/antisaccade latencies (in milliseconds) between the intranasal and oral oxytocin and placebo treatment conditions
Differential effects of intranasal and oral oxytocin administration on error rates of saccade/antisaccade for social (facial) versus non-social (shape) stimuli | 45 minutes - 100 minutes after treatment
  Comparison between social-specific error rates of saccade/antisaccade between the intranasal and oral oxytocin and placebo treatment conditions.

SECONDARY OUTCOMES:
Emotion-specific effects of intranasal and oral oxytocin administration on saccade/antisaccade latencies towards the separate facial emotions | 45 minutes - 100 minutes after treatment
  Comparison between emotion-specific saccade/antisaccade latencies (in milliseconds) between the intranasal and oral oxytocin and placebo treatment conditions
Emotion-specific effects of intranasal and oral oxytocin administration on saccade/antisaccade error rates for the separate facial emotions | 45 minutes - 100 minutes after treatment
  Comparison between emotion-specific saccade/antisaccade error rates between the intranasal and oral oxytocin and placebo treatment conditions

CONTACTS AND LOCATIONS:
Overall Officials: Keith Kendrick, PhD, Principal Investigator — University of Electronic Science and Technology of China (UESTC)
Locations (1):
- University of Electronic Science and Technology of China(UESTC), Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No